CLINICAL TRIAL: NCT02101528
Title: Determination of Muscle Strength in Parkinsonian Patients Through the Use of an Isokinetic Dynamometer
Acronym: CybexPD001
Status: Completed | Type: Observational
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Other Study IDs: CybexPD001; CybexPD001 (Other: Ospedale Generale di Zona "Moriggia-Pelascini")
Record Dates: First submitted 2014-03-21; First posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Parkinson's Disease
Keywords: Strength in PD patients; Isokinetic muscle strength
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PD Patients: PD patients with a diagnosis of "clinically probable" idiopathic PD in Hoehn-Yahr stage 2-3, with the ability to walk without any assistance, with mini-mental state examination score ≥26, without any relevant comorbidity or vestibular/visual dysfunctions limiting locomotion or balance.
- Controls: age and sex matched healthy volunteers

SUMMARY:
Decreased muscle strength has been reported to be a factor contributing to increased incidences of falling in the elderly patients causing fractures, joint dislocations, severe soft tissue lesions and head trauma. Parkinson's Disease (PD) patients often complain of weakness and it has been reported that they have reduced muscle strength, decreased rate of force development, impaired ability to maintain constant force, and increased muscle coactivation during balance perturbation tasks. The specific cause of this weakness is not known, and in this study the investigators have analyzed and measured isokinetic muscle strength in PD patients to clarify this issue. The investigators have compared the data obtained with those of age-matched controls.

DETAILED DESCRIPTION:
An isokinetic muscle action is defined by its performance at a constant speed or velocity. The laboratory measurements of isokinetic strength provides torque measurements throughout the active range of motion during a maximal effort. Torque is the force rotating about an axis and is produced and recorded from the angular motion. Consequently, the peak torque is an index of the muscular strength. Isokinetic testing was introduced as a quantitative measurement of both statistic and dynamic muscular contraction in which all variables involved (resistance, limb velocity, joint position) are under control. This is because isokinetic muscle testing allows objective, valid, and reliable measurement of the force produced by skeletal muscle during exercise at constant velocity and accommodating resistance and it is appropriate for measuring muscle strength and muscle endurance across the disability spectrum.

Decreased muscle strength has been reported to be a factor contributing to increased incidences of falling in the elderly patients causing fractures, joint dislocations, severe soft tissue lesions and head trauma. Parkinson's Disease (PD) patients often complain of weakness and it has been reported that they have reduced muscle strength, decreased rate of force development, impaired ability to maintain constant force, and increased muscle coactivation during balance perturbation tasks. The specific cause of this weakness is not known, and in this study the investigators have analyzed and measured isokinetic muscle strength in PD patients to clarify this issue. the investigators have compared the data obtained with those of age-matched controls.

ELIGIBILITY:
Inclusion Criteria:

* PD in stage 2-3 of Hoen&Yahr according to the United Kingdom Brain Bank criteria.

Exclusion Criteria:

* Atypical parkinsonisms
* PD patients with relevant orthopedic
* Rheumatic and muscular conditions

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with PD in stage 2-3 of Hoen&Yahr according to the United Kingdom Brain Bank criteria.
  Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Isokinetic strength | One month
  Laboratory measurements of isokinetic strength

SECONDARY OUTCOMES:
Muscle functionality | One month
  To establish whether a Intensive Rehabilitation Treatment change the muscle functionality in these patients, and to determine whether isokinetic dynamometry is a reliable method for evaluating muscle strength in patients with PD.
  Muscle strength was measured in lower limbs with the subjects in a sitting position with hip flexed at 90°. To account for the influence of the gravity effect torque, data were corrected by the weight of the subject's lower limb at 45°. Subjects were tested at three fixed angular velocities: 90°/s, 120°/s, 180°/s. The subjects began each isokinetic contraction with the knee flexed at 90° and continued through the full range of motion. Peaks torque were obtained from the maximum isokinetic tests and subsequently analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Principal Investigator — Ospedale Generale di Zona "Moriggia-Pelascini", Gravedona ed Uniti (CO), Italy
Locations (1):
- Fondazione Salvatore Maugeri, Montescano, Pavia, Italy